CLINICAL TRIAL: NCT01575964
Title: Biomechanical Assessment of Femoroacetabular Impingement
Acronym: FAI
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Andrew Anderson, Associate Professor, University of Utah
Other Study IDs: 51053
Record Dates: First submitted 2012-03-06; First posted 2012-04-12 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Femoro Acetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the influence of FAI abnormalities on hip joint biomechanics.

DETAILED DESCRIPTION:
The purpose of this study is to quantify hip biomechanics of subjects with and without FAI.

The results of this study will advance our understanding of how the FAI alters the biomechanics of the hip joint, improving diagnosis and directing treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with hip pain subsequently diagnosed as femoroacetabular impingement
* Subjects who meet the following radiographic criterion of cam or pincer FAI, will be given the opportunity to volunteer in this study.
* Subjects that demonstrate a cross-over-sign or a lateral center edge angle (LCEA) without an alpha angle, will be classified as having pincer FAI.
* Subjects with an alpha angle, without a cross-over sign or LCEA, will be categorized as having cam type FAI.
* Finally, with at least one cam (alpha angle) and pincer sign "cross-over-sign or a lateral center edge angle (LCEA)" will be classified as mixed FAI.

Control Population Inclusion Criteria:

* 12 controls will consist of volunteers in the same age range as the subject groups (18-35 years).
* Control hips will be screened with a standard AP radiograph. Normal volunteers who have radiographic evidence of FAI, dysplasia or other joint deformities will be excluded.

Exclusion Criteria:

* Subjects who have radiographic evidence of osteoarthritis (Tonnis Grade III or IV) will be excluded as this study focuses on the mechanics of hips before prominent cartilage damage.
* Subjects who have had prior procedures to correct FAI or other hip conditions will be excluded (exploratory procedures will be included).
* Minors (under age 18), mentally disabled, persons incarcerated, on parole, probation awaiting trial, or pregnant women are excluded from this study.
* A human Chorionic Gondaotropin (hCG) urine pregnancy test will be performed on all women prior to the study.
* To limit the annual radiation exposure to any participating volunteers, we will exclude anyone who has had a CT scan or participated in a research study involving ionizing radiation in the past 12 months.

Motion Capture Exclusion Criteria:

* Subjects who are unwilling or unable to perform the proposed activities of daily living or undergo the clinical exams will be dismissed.
* Subjects with a BMI less than 30 (www.nhlbisupport.com/bmi/) or those with dense hip musculature/wide hips (maximum of 42 cm of circumferential hip length) will be excluded.

CT Exclusion Criteria:

* Subjects who are unwilling or unable to remain still.
* Subjects who are allergic to contrast agent and/or lidocaine will be dismissed.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal subjects and subjects with femoroacetabular impingement.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2012-01; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Data Collection | Follow-up Visit
  We will calculate hip joint kinematics. Statistical analysis of the results will allow comparisons between normal and FAI subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Anderson, Principal Investigator — Orthopedic Surgery Operations
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States